CLINICAL TRIAL: NCT00320840
Title: The Contribution of Internal and Familial Resources to the Development of Motherhood. Long Term Follow Up of Mothers With Twins and Preterm Infants Versus Mothers With Single Full Term Infants
Brief Title: Internal and Familial Resources and Motherhood. Follow Up of Mothers With Twins and Preterm Infants Versus Mothers With Single Full Term Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4131-JK-CTIL
Record Dates: First submitted 2006-04-30; First posted 2006-05-03 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-04

CONDITIONS: Twins; Preterm Infants
Keywords: preterm infants; twins; motherhood; internal resources; familial resources

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
To evaluate the contribution of internal and familial resources on the development of motherhood in a population of mothers having preterm twin infants and comparing this population to a population of mothers giving birth to single (or twins) full term infants.

DETAILED DESCRIPTION:
150 mothers will participate in this study. The study is using 4 questionnaires at infants ages of 1 month, 1 year, 2 years and 4 years. The questionnaires are involving communication skills,grandparents support, stress feelings, psychological parameters, parity functioning, infant temperament, self assessment, maternal and infant medical background and twins and brotherhood evaluation.

a comparison will be done between mothers to preterm twins and mothers to single full term infants.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants
* twins

Exclusion Criteria:

-

Ages: 2 Weeks to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 2006-05; Study Completion 2012-05

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kuint, MD, Study Director — Sheba Medical Center
Locations (1):
- Sheba medical center - Neonatal Department, Ramat Gan, Israel